CLINICAL TRIAL: NCT01708824
Title: The Acceptability and Feasibility of a Diet and Physical Activity Intervention to Prevent Recurrence in Colorectal Cancer Survivors: a Phase 2 Study
Brief Title: Diet and Physical Activity Intervention in CRC Survivors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: World Cancer Research Fund International (Other)
Responsible Party: Principal Investigator, Dr. Judy Wai-Chu Ho, Consultant, Honorary Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: WCRF 2012/595
Record Dates: First submitted 2012-10-11; First posted 2012-10-17 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; cancer survivor; western pattern diet; physical activity; behavioral intervention; acceptability; feasibility; randomized controlled trial; compliance
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity; Patient Compliance | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- dietary (Experimental): Dietary intervention to meet the target of
  1.<5 servings of red/processed meat weekly; <2 servings would be processed meat 2.2 servings of refined grains daily
  Interventions: Behavioral: Dietary
- physical activity (Experimental): Physical activity intervention with the following targets:
  1. General health target - 30 minutes of moderate-to-vigorous physical activity (MVPA) 5 days per week (i.e. 10 MET-hours/week);
  2. Cancer outcome target - 60 minutes of MVPA 5 days per week (i.e. 18-20 MET-hours/week)
  Interventions: Behavioral: Physical activity
- dietary and physical activity (Experimental): Meeting both the dietary and physical activity targets
  Interventions: Behavioral: Dietary; Behavioral: Physical activity
- usual care (No Intervention): Follow the general lifestyle advice in accordance with the recommendations of the Department of Health in Hong Kong available in the public domain

INTERVENTIONS:
Behavioral: Dietary — Dietary intervention to meet the target of
  1. <5 servings of red/processed meat weekly; <2 servings would be processed meat
  2. 2 servings of refined grains daily
  Arms: dietary; dietary and physical activity
Behavioral: Physical activity — Physical activity intervention with the following targets:
  1. General health target - 30 minutes of moderate-to-vigorous physical activity (MVPA) 5 days per week (i.e. 10 MET-hours/week);
  2. Cancer outcome target - 60 minutes of MVPA 5 days per week (i.e. 18-20 MET-hours/week)
  Arms: dietary and physical activity; physical activity

SUMMARY:
Background - Colorectal cancer (CRC) incidence is increasing at an alarming rate in Hong Kong. A recent report concluded physical activity (PA) protects against colon cancer and foods low in dietary fibre, red meat and processed meat cause CRC. Yet, the influence of lifestyle factors on cancer outcome (i.e. recurrence and survival rates) in CRC survivors is largely unknown.

Objectives & hypothesis - Our study aims to evaluate the acceptability of two behavioural interventions for CRC survivors intended to improve cancer outcome and designed to (1) increase PA levels and (2) reduce consumption of a Western diet.

The investigators hypothesize that the proposed interventions are (1) efficacious in changing the two targeted behaviours; and (2) acceptable to CRC survivors.

Settings and methods - Phase 2 feasibility trial. Two hundred and twenty-four CRC survivors within 12 months of completion of cancer treatment and without evidence of persistent/recurrent disease will be recruited from four public hospitals in Hong Kong after informed consent. Subjects will be randomized in a 2x2 factorial design for the two targeted behaviours prescribed over 12 months. Primary outcome measure is whether the target levels of PA and dietary intake could be met at the end of intervention. Secondary outcome measures include: (1) magnitude of changes in PA level and dietary intakes; (2) rates and determinants of compliance; (3) facilitators and barriers to behavioural change; (4) measurement of theoretical constructs underlying PA and dietary interventions; (5) possible health benefits and side effects (PA-associated injury and nutritional deficiency) arising from the interventions. Outcome will be assessed at baseline, 6 months into intervention and then at 0, 6 and 12 months post-intervention.

Impact - If proven feasible, our intervention programme would pave way for a large randomized controlled trial testing the effect of PA and diet on the treatment outcome of CRC.

DETAILED DESCRIPTION:
Background - Colorectal cancer (CRC) incidence is increasing at an alarming rate in Hong Kong. A recent World Cancer Research Fund (WCRF) report concluded physical activity (PA) protects against colon cancer and foods low in dietary fibre, red meat and processed meat cause CRC. Yet, the influence of lifestyle factors on cancer outcome (i.e. recurrence and survival rates) in CRC survivors is largely unknown. Our literature review showed a paucity of published studies on lifestyle intervention in CRC survivors; none had investigated the effect of such intervention on cancer outcomes.

With advances in treatment, CRC survivors live longer. Many of them are motivated to make lifestyle changes. However, our qualitative research has shown a huge service gap in the provision of appropriate PA and dietary advice to CRC survivors. Many patients were unaware of the link between PA and diet with CRC outcome but most demonstrated acceptance of lifestyle intervention. Yet, there is currently no scientifically-based evidence to allow firm recommendations to be made.

Objectives & hypothesis - Our study aims to evaluate the acceptability of two behavioural interventions for CRC survivors intended to improve cancer outcome and designed to (1) increase PA levels (to 60 minutes of moderate PA 5 days/week) and (2) reduce consumption of a Western diet (<5 servings of red/processed meat weekly and 2 servings of refined grain daily).

We hypothesize that the proposed interventions are (1) efficacious in changing the two targeted behaviours; and (2) acceptable to CRC survivors with compliance rates of about 80%.

Settings and methods - The study follows the Medical Research Council Framework for the design and evaluation of complex interventions. Phases 0 and 1 (funded by WCRF) have been completed.

This application seeks funding for a Phase 2 feasibility trial. Two hundred and twenty-four CRC survivors within 12 months of completion of cancer treatment and without evidence of persistent/recurrent disease will be recruited from four public hospitals in Hong Kong after informed consent. Subjects will be randomized in a 2x2 factorial design for the two targeted behaviours prescribed over 12 months. Primary outcome measure is whether the target levels of PA and dietary intake could be met at the end of intervention. Secondary outcome measures include: (1) magnitude of changes in PA level and dietary intakes; (2) rates and determinants of compliance by questionnaire; (3) facilitators and barriers to behavioural change by questionnaire; (4) measurement of theoretical constructs underlying PA and dietary interventions by questionnaire; (5) possible health benefits (body composition, physical fitness, quality of life and mood) and side effects (PA-associated injury and nutritional deficiency) arising from the interventions. Outcome will be assessed at baseline, 6 months into intervention and then at 0, 6 and 12 months post-intervention (i.e. at baseline, 6, 12, 18 and 24 months after the start of intervention).

Impact - To the best of our knowledge, this is the first behavioural intervention model targeting PA and reduced consumption of a Western diet in CRC survivors. If proven feasible, our intervention programme would pave way for a large randomized controlled trial testing the effect of PA and diet on the treatment outcome of CRC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven colorectal adenocarcinoma;
2. Within one year of completion of main cancer treatment

Exclusion Criteria:

1. Persistent/recurrent disease upon recruitment;
2. Current cancer treatment;
3. Hereditary CRC syndromes;
4. Known contraindication to PA;
5. Illiteracy;
6. Weekly red/processed meat < 5 servings and daily refined grains < 2 servings
7. Weekly MPA > 300 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Whether the PA and dietary intake targets are met at the end of intervention; | at the end of 12 months of intervention
  Whether the PA and dietary intake targets are met at the end of intervention; i.e.
  1. PA group: achieve PA targets or not
  2. Dietary group: achieve dietary target or not
  3. PA + dietary group: achieve both PA and dietary targets or not
  4. Control group: achieve PA or dietary target or not

SECONDARY OUTCOMES:
Magnitude of change in PA level using objective accelerometry | 6, 12, 18 and 24 months after start of intervention (i.e. interim, 0, 6 and 12 months post-intervention)
Magnitude of change in each component of dietary target using validated food frequency questionnaire (FFQ); | 6, 12, 18 and 24 months after start of intervention (i.e. interim, 0, 6 and 12 months post-intervention)
Rate and determinants of compliance with intervention; | at the end of 12 months of intervention
  Rates of compliance - measured by rate of completion of assignment; determinants of compliance measured by a questionnaire
Facilitators and barriers to intervention | at the end of intervention
  Measured by (a) qualitatively during the last group meeting and (b) quantitatively by questionnaire
Measurement of theoretical constructs underlying PA and dietary interventions | 6, 12, 18 and 24 months after start of intervention (i.e. interim, 0, 6 and 12 months post-intervention)
  Using questionnaire specifically desinged to measure these theoretical constructs
Other possible health benefits arising from the intervention | at 12 and 24 months after start of intervention (i.e. at 0 and 12 months post-intervention)
  including
  1. Changes in body composition via body mass index (BMI)
  2. Changes in body fat and/or visceral fat via waist-hip ratio (WHR) and bioelectrical impedance analysis
  3. Physical fitness in the form of submaximal oxygen uptake as predicted by 6-minute ergometry
  4. Quality-of-life/mood via validated tools (SF12, FACT, HADS and PSS);
Possible side effects arising from the intervention | at 6, 12, 18 and 24 months after start of intervention (i.e. interim, 0, 6 and 12 months post-intervention)
  including
  1. PA-associated injury
  2. Dietary deficiency - (i) anaemia (haemoglobin level); (ii) energy and protein deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Judy WC Ho, MBBS, Principal Investigator — Queen Mary Hospital, University of Hong Kong
Locations (4):
- China (4):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Yan Chai Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No
no consent has been obtained to make individual participant data available

REFERENCES:
- [Derived] Wong JYH, Ho JWC, Lee AM, Fong DYT, Chu N, Leung S, Chan YYW, Lam SH, Leung IPF, Macfarlane D, Cerin E, Taylor AJ, Cheng KK. Lived experience of dietary change among Chinese colorectal cancer survivors in Hong Kong: A qualitative study. BMJ Open. 2021 Aug 25;11(8):e051052. doi: 10.1136/bmjopen-2021-051052. PMID 34433608
- [Derived] Ho M, Ho JWC, Fong DYT, Lee CF, Macfarlane DJ, Cerin E, Lee AM, Leung S, Chan WYY, Leung IPF, Lam SHS, Chu N, Taylor AJ, Cheng KK. Effects of dietary and physical activity interventions on generic and cancer-specific health-related quality of life, anxiety, and depression in colorectal cancer survivors: a randomized controlled trial. J Cancer Surviv. 2020 Aug;14(4):424-433. doi: 10.1007/s11764-020-00864-0. Epub 2020 Feb 18. PMID 32072434
- [Derived] Ho JW, Lee AM, Macfarlane DJ, Fong DY, Leung S, Cerin E, Chan WY, Leung IP, Lam SH, Taylor AJ, Cheng KK. Study protocol for "Moving Bright, Eating Smart"- A phase 2 clinical trial on the acceptability and feasibility of a diet and physical activity intervention to prevent recurrence in colorectal cancer survivors. BMC Public Health. 2013 May 20;13:487. doi: 10.1186/1471-2458-13-487. PMID 23688320